CLINICAL TRIAL: NCT05856643
Title: Single-arm, Open-label Clinical Study of SZ011 in the Treatment of Ovarian Epithelial
Brief Title: Single-arm, Open-label Clinical Study of SZ011 in the Treatment of Ovarian Epithelial Carcinoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shantou University Medical College (Other)
Collaborators: Guangdong ProCapZoom Biosciences Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Li Congzhu, Chief physician, Shantou University Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCZCTP-230316-002
Record Dates: First submitted 2023-05-03; First posted 2023-05-12 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Ovarian Epithelial Carcinoma
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SZ011 CAR-NK (Experimental)
  Interventions: Drug: SZ011 CAR-NK

INTERVENTIONS:
Drug: SZ011 CAR-NK — In the escalation study, the minimum initial dose was 5.0×10^6 cells, then increased to 1.0×10^8, 2.0×10^8and 5.0×10^8 cells. The infusion is given every 2 weeks.

SUMMARY:
This study was a single-center, open-label, investigator-initiated clinical trial (IIT) to observe and investigate the clinical safety and efficacy of SZ011 in the treatment of ovarian epithelial carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 18-80;
2. Histologically confirmed ovarian epithelial carcinoma;
3. Ovarian cancer patients who have failed or relapsed after first-line treatment, with or without other treatments;
4. At least one measurable lesion according to RECIST 1.1 ;
5. Positive expression of mesothelin in ovarian cancer tumors;
6. Functional status score (KPS) ≥80;
7. Expected survival ≥28 weeks;
8. The function of important organs meets the following requirements: absolute neutrophil count ≥1.5×109/L; platelets count ≥50×109/L; hemoglobin ≥80g/L; serum albumin ≥2.5g/dL; bilirubin ≤1.5 times ULN; ALT and AST ≤3 times ULN; serum creatinine ≤1.5 times ULN;
9. Able to understand the informed consent form, voluntarily participate, and sign the informed consent form;
10. The subject or their partner agrees to take the contraceptive measures recognized by the trial within 1 month after signing the informed consent form until the end of the study.

Exclusion Criteria:

1. Exclusion criteria include those who have had other malignant tumors within the past 5 years, except for those who have been cured of basal cell carcinoma, cervical carcinoma in situ, and breast cancer that has not recurred for >3 years after radical surgery.
2. Patients known to have central nervous system metastasis or leptomeningeal disease are excluded.
3. Patients who have experienced arterial thromboembolic events (including myocardial infarction, cardiac arrest, cerebrovascular accident, ischemic stroke, deep venous thrombosis of CTCAE 5.0 grade ≥3) or a history of pulmonary embolism within 6 months prior to enrollment are excluded.
4. Patients with a history of serious bleeding disorder within 6 months prior to screening, or those with a clear tendency to bleed (such as esophageal varices at risk of bleeding, active ulcer lesions, fecal occult blood >2+) as judged by the investigator, are excluded.
5. Patients with congenital or acquired immunodeficiency (such as HIV infection), active hepatitis B or C virus infection, or other severe infectious diseases are excluded.
6. Patients with clinically significant cardiovascular disease:

   1. Uncontrolled hypertension (systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥110mmHg) despite treatment;
   2. History of myocardial infarction or unstable angina pectoris within 6 months prior to enrollment;
   3. Congestive heart failure or NYHA class II heart failure;
   4. Severe symptomatic arrhythmia requiring medication, excluding asymptomatic atrial fibrillation that is controllable.
7. Pregnant or lactating women are excluded.
8. Those who have participated in or are currently participating in other clinical trials within the past three months are excluded.
9. Patients considered unsuitable for this clinical trial by the investigator are excluded.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-08-13 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events (AEs) | Up to 6 months after infusion
  To evaluate the safety of SZ011 CAR-NK Cells
Objective response rate (ORR) | Up to 6 months after infusion
  To evaluate the ORR of SZ011 CAR-NK Cells
Overall survival (OS) | Up to 6 months after infusion
  To determine the anti-tumor effectivity of SZ011 CAR-NK Cells
Progression-free survival (PFS) | Up to 6 months after infusion
  To determine the anti-tumor effectivity of SZ011 CAR-NK Cells

CONTACTS AND LOCATIONS:
Locations (1):
- Shantou University Medical College, Shantou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No